CLINICAL TRIAL: NCT00010738
Title: Effects of Meditation on Mechanism of Coronary Heart Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: R01 AT000226-01M; R01AT000226-01 (NIH); NCT00009399 (obsolete NCT alias)
Record Dates: First submitted 2001-02-02; First posted 2001-02-05 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-07

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease | interventions — Meditation

INTERVENTIONS:
Procedure: Meditation

SUMMARY:
To study the effects of Transcendental Meditation on Coronary Heart Disease

DETAILED DESCRIPTION:
Recent advances in our understanding of the pathophysiology of acute cardiac events - specifically, identification of the roles that arterial vasomotor dysfunction and autonomic nervous system imbalances play in the pathophysiologic cascade during such acute events - provides a platform for new mechanistic investigation of the interplay of psychosomatic stress and CHD (coronary heart disease). Preliminary evidence further suggests that Complementary and Alternative Medicine (CAM) practices, such as the Transcendental Meditation (TM) technique, can not only reduce stress but also reduce acute cardiac events in patients with CHD. Based on these and related data, we propose a randomized, blinded, controlled study of the effects of one CAM practice, the TM technique, compared to a control group, on the primary outcomes of (1) arterial vasomotor dysfunction (brachial artery reactivity); (2) autonomic nervous system imbalances (heart rate variability); (3) transient myocardial ischemia (ST-segment depression); and (4) the secondary outcomes of psychological stress and quality of life (anger, hostility, anxiety, depression, perceived health, disease-specific symptoms, and life stress/social resources).

ELIGIBILITY:
Inclusion Criteria:

* Able to attend training sessions and meetings
* Local residence

Exclusion Criteria:

* Comorbid disease precluding survival in group
* MI, unstable angina, CABG or PTCA within last three months.
* Cognitive/psychological/substance abuse impairment
* Atrial fibrillation, predominant pacemaker rhythm or significant conduction system disease
* Significant valvular heart disease
* Class III or IV heart failure
* Renal failure
* Participating in a formal stress management program
* Participation in another trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145
Dates: Start 1999-09; Study Completion 2002-08

CONTACTS AND LOCATIONS:
Overall Officials: C. Noel Bairey Merz, M.D., Principal Investigator — Preventive and Rehabilitative Cardiac Center
Locations (1):
- Preventive and Rehabilitative Cardiac Center, Los Angeles, California, United States